CLINICAL TRIAL: NCT05777330
Title: Continuous Monitoring of Glycemic Variability to Predict Dys- and Hyperglycemia in Asymptomatic Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Breakthrough T1D (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PredicT1D
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — Glucose Tolerance Test; Glucose Clamp Technique; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Autoantibody-positive individuals (Other)
  Interventions: Diagnostic Test: Oral glucose tolerance test (OGTT); Diagnostic Test: Hyperglycemic clamp test; Diagnostic Test: Continuous glucose monitoring

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test (OGTT) — Longitudinal study using repeated OGTT, CGM and hyperglycemic clamp tests to evaluate glycemic variability, beta cell function and insulin action in individuals at moderate, high and very high risk of clinical onset of type 1 diabetes.
  OGTT is performed every 6 months (every 3 months in case of dysglycemia) in all participants.
  Other Names: OGTT
Diagnostic Test: Hyperglycemic clamp test — Longitudinal study using repeated OGTT, CGM and hyperglycemic clamp tests to evaluate glycemic variability, beta cell function and insulin action in individuals at moderate, high and very high risk of clinical onset of type 1 diabetes.
  Clamp test is performed every 12 months in single autoantibody-positive participants and every 6 months in multiple autoantibody-positive participants. Clamp tests are not performed in participants aged between 5-11 years.
  Other Names: clamp
Diagnostic Test: Continuous glucose monitoring — Longitudinal study using repeated OGTT, CGM and hyperglycemic clamp tests to evaluate glycemic variability, beta cell function and insulin action in individuals at moderate, high and very high risk of clinical onset of type 1 diabetes.
  A 10-day CGM recording is performed every 6 months (every 3 months in case of dysglycemia) in all participants.
  Other Names: Dexcom G6; CGM

SUMMARY:
The goal of this longitudinal clinical trial is to measure variability of interstitial glucose levels with a user-friendly real-time continuous glucose monitoring (CGM) technology at regular intervals in normo- and dysglycemic multiple autoantibody-positive individuals (age 5-39 years), in comparison with single autoantibody-positive individuals in the same age range. Participants will asked to undergo repeated oral glucose tolerance tests (OGTTs) (age 5-39 years) and hyperglycemic clamp tests (age 12-39 years) in parallel for a period of at least 2-3 years. In case of confirmed dysglycemia, we propose to perform CGM and OGTT every 3 months.

The main questions the study aims to answer are:

1. Do the amplitude and time trends of CGM-derived glycemic variability indices and OGTT- and clamp-derived variables differ between the intermediate, high and very high risk groups?
2. Can (changes in) CGM-derived glycemic variability indices predict/detect dysglycemia in initially normoglycemic (single or multiple autoantibody-positive) individuals with the same diagnostic efficiency as OGTT- or clamp-derived variables?
3. Can (changes in) CGM-derived glycemic variability indices predict clinical onset in (stage 1 or 2) multiple autoantibody-positive individuals with the same diagnostic efficiency as OGTT- or clamp-derived variables?
4. Can correlating (changes in) CGM-derived indices with (changes in) OGTT- and clamp-derived variables help to better understand the sequence of events leading to dysglycemia and clinical onset, as well as the relative contribution of beta cell function and insulin action to glycemic variability according to disease stage and biological and phenotypical characteristics of the individuals?

DETAILED DESCRIPTION:
Type 1 diabetes is a for now incurable disease caused by a major immune-mediated loss of insulin-producing pancreatic beta cells, can lead to potentially severe acute and chronic complications and requires a lifelong insulin treatment. Clinical onset of type 1 diabetes is preceded by an asymptomatic disease phase of highly variable duration, which is signaled by the presence of multiple (≥2) types of islet autoantibodies. Multiple autoantibody-positive individuals, with blood glucose levels still within normal limits (defined as stage 1 type 1 diabetes) have a 90% risk of developing symptomatic disease within the next 20 years. The development of dysglycemia (stage 2 type 1 diabetes) - i.e. disturbed blood glucose levels during an oral glucose tolerance test (OGTT) - dramatically raises the risk of impending clinical onset to 90% within 5 years. Identifying individuals at high risk of impending clinical onset of type 1 diabetes is important for early diagnosis, for reducing the incidence of inaugural ketoacidosis, and for enrolling participants of choice in immune intervention trials before and at clinical diagnosis, aiming to develop an effective cure or even better, prevention. The hyperglycemic clamp test is the gold standard for assessing beta cell function and has also been validated for estimating insulin action in parallel. Decreased clamp-derived measures of islet function and insulin action have been shown to outperform OGTT-derived variables for predicting progression to symptomatic disease. However, the repeated performance of both OGTTs and clamps are cumbersome and difficult to implement on a large scale in a seemingly healthy population. In contrast, continuous glucose monitoring (CGM) methods nowadays avoid the need of frequent calibration based on capillary blood measurements obtained by finger pricks. They also allow to detect more subtle glycemic fluctuations over longer observation periods and on a more frequent basis than achievable with OGTT, and to derive a wide variety of indices of glycemic variability. Preliminary findings suggest that repeated CGM metrics in stage 1 asymptomatic diabetes could represent a minimally invasive alternative to OGTT for early detection or prediction of stage 2 asymptomatic disease, provided that increased CGM-derived glycemic excursions can be shown to coincide with or precede OGTT-inferred dysglycemia, respectively, in a longitudinal study. In addition, it is anticipated that further increasing glycemic excursions may forecast impending clinical onset. Using the capacity of the nationwide network of the Belgian Diabetes Registry, we therefore propose a longitudinal study to measure variability of interstitial glucose levels with a userfriendly real-time CGM technology at regular intervals (every 6 months) during follow-up of multiple autoantibody-positive first-degree individuals (age 5-39 years; n>50) of type 1 diabetes patients, in comparison with single autoantibody-positive individuals (n>25). In parallel repeated OGTTs (age 5-39 years) and hyperglycemic clamp tests (age 12-39 years) will be performed for a period of at least 2-3 years. We anticipate that, especially when using up-to-date CGM technology, (i) the amplitude and time trends of various glycemic variability indices - alone or in combination - will differ between groups of individuals at moderate (single autoantibody-positive), high (stage 1), and very high (stage 2) risk of impending clinical onset (stage 3); (ii) (changes in) CGM-derived glycemic variability indices will be able to predict and/or diagnose stage 2 asymptomatic type 1 diabetes and clinical onset (stage 3) with a diagnostic efficiency equaling that of variables derived from (repeated) OGTT or clamp tests; (iii) correlating CGM metrics with hyperglycemic clamp- and OGTT-derived indices of beta cell function and insulin action will help to understand the relative contribution of both components to disease progression in general, and to glycemic variability in particular.

ELIGIBILITY:
Inclusion Criteria:

1. aged 5-39 years at inclusion;
2. absence of diabetes meeting the clinical diagnostic American Diabetes Association (ADA) criteria;
3. persistently positive for one or multiple types of autoantibodies among IAA, GADA, IA-2A and ZnT8A.

Exclusion Criteria:

1. Pregnancy or lactation in women; <6 months postpartum
2. Diabetes meeting the clinical diagnostic ADA criteria;
3. Use of illicit drugs, or overconsumption of alcohol, or history of drug or alcohol abuse;
4. Being legally incapacitated, having significant emotional problems at the time of the study, or having a history of psychiatric disorders;
5. Treatment with immune modulating or diabetogenic medication (e.g. corticosteroids) or medication that act to lower glycemia (oral antidiabetics) or agents that may influence insulin sensitivity or secretion;
6. Gastric bypass or banding;
7. History of acute or chronic pancreatitis, or (partial) pancreatectomy
8. History of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risks to the subjects.

Ages: 5 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Progression to persistent dysglycemia | 2-3 years
  In initially normoglycemic (single or multiple) autoantibody-positive individuals
Progression to persistent dysglycemia and stage 3 type 1 diabetes | 2-3 years
  In all multiple autoantibody-positive individuals

CONTACTS AND LOCATIONS:
Overall Officials: Bart Keymeulen, Principal Investigator — Vrije Universiteit Brussel
Locations (6):
- Belgium (6):
  - Clinique CHC MontLégia, Liège, Liège
  - A.Z. Sint-Jan Brugge, Bruges, West-Vlaanderen
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - Universitair Ziekenhuis Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No
We opt to restrict data access as the project involves personal and sensitive data.
  A specific data use agreement could be considered for data sharing after the end of the project.